CLINICAL TRIAL: NCT06706882
Title: The Role of Executive Functioning in Complex Post-Traumatic Stress Disorder Among Female Survivors of Intimate Partner Violence (BELIEVE-CPTSD)
Brief Title: The Role of Executive Functioning in Complex Post-Traumatic Stress Disorder Among Female Survivors of Intimate Partner Violence
Acronym: BELIEVE-CPTSD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Natalia Hidalgo Ruzzante, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2022-143060NB-I00; PID2022-143060NB-I00 (Other: Ministry of Science and Innovation)
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Neuropsychological Rehabilitation Program (VIRTRAEL/LUCCIDY); Standard Training (TAU)
Keywords: Intimate partner violence; Posttraumatic Stress Disorder; Complex Postrraumatic Stress Disorder; Neuropsychological functioning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel group randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Training: VIRTRAEL/LUCCIDY (Experimental): The neuropsychological rehabilitation program VIRTRAEL/LUCCIDY is designed for cognitive assessment and stimulation, shown to improve verbal learning, memory, attention, reasoning, and planning. It consists of 11 exercises over 9 sessions, each lasting 60 minutes. The platform adapts the difficulty of exercises based on performance through an algorithm, focusing on cognitive functions like attention, memory, and planning. To maintain motivation, the program includes varied exercises, avatars, and rewards. The exercises are ecologically designed to simulate daily activities for real-life application. Sessions involve tasks like shopping lists, puzzles, and memory challenges. Link: http://www.everyware.es/webs/virtrael/#home
  Interventions: Behavioral: Experimental Training: VIRTRAEL/LUCCIDY
- Standard Training: Reflection Group (TAU) (Active Comparator): It is a group work offered to survivor women of IPV in municipal and provincial centers (CIMs) of the Women's Institute. The objective of this intervention is to provide women with a space for group reflection, as well as a series of skills and tools. Concrete topics are presented, including those related to intervention in crisis situations from a gender perspective. It lasts for 9 sessions (60 minutes per session) with a frequency of one session per week.
  The sessions cover themes such as the idealization of women as caregivers (Session 1), gender conflicts (Session 2), guilt when deviating from gender expectations (Session 3), dependence on others for self-worth (Session 4), and romantic love as a tool to fulfill men's needs over women's (Session 5). They explore intimate partner violence (IPV) as a conflict strategy (Session 6), family's role in socialization (Session 7), fears of abandonment (Session 8), and life skills for independence (Session 9).
  Interventions: Behavioral: Active Comparator: Standard Training: Reflection Group (TAU) (Andalusian Institute of Women, 2010)

INTERVENTIONS:
Behavioral: Experimental Training: VIRTRAEL/LUCCIDY — Cognitive stimulation of the different cognitive functions to be addressed will be conducted in the following sessions:
  * Session 1: Shopping lists. Balls. Gift shopping. Long-term memory of the Shopping List.
  * Session 2: Disordered objects. Whats different? Semantic series. Logical series. Puzzle pieces. Semantic analogies.
  * Session 3: Classifiable objects. Gift shopping. Bag of objects.
  * Session 4: Shopping lists. Balls. Disordered objects. Long-term memory of the Shopping List.
  * Session 5: Semantic series. Logical series. Puzzle pieces. Semantic analogies. Gift shopping.
  * Session 6: Classifiable objects. Bag of objects. Disordered objects.
  * Session 7: Shopping lists. Semantic series. Logical series. Puzzle pieces. What's different? Semantic analogies. Long-term memory of the Shopping List.
  * Session 8: Disordered objects. Gift shopping. Balls.
  * Session 9: Bag of objects. Semantic series. Logical series. Whats different? Semantic analogies. Classifiable objects.
  Arms: Experimental Training: VIRTRAEL/LUCCIDY
Behavioral: Active Comparator: Standard Training: Reflection Group (TAU) (Andalusian Institute of Women, 2010) — This 9-session program explores how societal norms shape women's roles and identities. In Session 1, it discusses how women are socially positioned as caretakers in relationships and introduces the concept of the self in relation. Session 2 delves into gender conflicts, focusing on the tension between societal demands and personal desires. Session 3 explores guilt when women fail to meet expected roles, and the fear of being selfish when prioritizing their own needs. Session 4 examines how dependence is fostered by seeking external validation for self-worth. Session 5 critiques romantic love as a cultural tool to prioritize men desires over women. Session 6 analyzes how intimate partner violence (IPV) emerges as a means to maintain power imbalances in relationships. Session 7 looks at the family role in socializing women, while Session 8 explores fears of abandonment. Finally, Session 9 focuses on building life skills and concludes the program.
  Arms: Standard Training: Reflection Group (TAU)

SUMMARY:
This project aims to investigate neuropsychological alterations in women with PTSD (Post-Traumatic Stress Disorder) and complex PTSD (CPTSD), survivors of intimate partner violence (IPV), and to implement a cognitive stimulation program. The specific objectives are:

* To establish the prevalence and severity of neuropsychological alterations in women victims of IPV and to define their profile according to the type of violence suffered.
* To analyze the differences in neuropsychological alterations between PTSD and CPTSD.
* To implement a cognitive stimulation program in women with CPTSD.
* To evaluate whether this program reduces symptoms of DSO (Disorders of Extreme Stress Not Otherwise Specified) and classic post-traumatic symptoms.
* The hypotheses suggest that women victims of IPV will present lower scores in executive functions, attention, and memory, a higher prevalence of CPTSD, and that the cognitive stimulation program will improve complex post-traumatic sequelae.

Methodology: Women victims of IPV attended at the CIMs of Andalusia will be randomly selected, with support from with support from the Andalusian Women Institute. Participants: 100 women victims of IPV and 100 non-victims. Inclusion criteria are literacy and, for IPV, having experienced partner violence. Those with a history of brain damage, previous psychopathological alterations, or diseases affecting cognition will be excluded. Evaluation: It will include sociodemographic surveys, violence assessment, psychopathological alterations, DSO symptoms, and neuropsychological assessments. Intervention: A cognitive stimulation program (VIRTRAEL/LUCCIDY) and a standard training (Reflection Group; TAU) in groups. Nine weekly sessions will be conducted, evaluating pre- and post-treatment and follow-up at 3 months.

DETAILED DESCRIPTION:
STARTING HYPOTHESIS AND OBJECTIVES We hypothesize that women who have experienced IPV will demonstrate lower scores on standardized neuropsychological tests, particularly in executive functions, attention, and memory, as well as a higher prevalence of a diagnosis of C-PTSD (Complex Post-Traumatic Stress Disorder) compared to non-victimized women. Furthermore, these neuropsychological alterations are expected to be more closely associated with specific symptoms of C-PTSD than with those of PTSD. Therefore, we hypothesize that the implementation of a cognitive stimulation program will more effectively improve complex post-traumatic sequelae than classic symptoms.

General Objective: The general objective of this project is to study the mediating role of neuropsychological alterations in PTSD and C-PTSD (according to ICD-11 diagnostic criteria) in women survivors of IPV and to implement a neuropsychological rehabilitation program.

Specific Objectives:

1. To establish the prevalence and severity of alterations in neuropsychological functioning in women survivor of IPV, as well as to define the profile of neuropsychological sequelae, and differentiate it according to the type of violence experienced (psychological, physical, and sexual).
2. To analyze differences in neuropsychological alterations between Post-Traumatic Stress Disorder and Complex Post-Traumatic Stress Disorder.
3. To implement a neuropsychological rehabilitation program (VIRTRAEL-LUCCIDY) in women survivors of IPV.
4. To examine whether the application of a neuropsychological rehabilitation program reduces DSO symptoms (negative self-concept, difficulties in emotional regulation, and difficulties in interpersonal relationships) in survivor women, as well as classic Post-Traumatic Symptoms.

Specific Hypotheses:

1. Women who have experienced IPV will demonstrate lower scores on standardized neuropsychological tests, particularly in executive functions, attention, and memory, compared to non-victimized women.
2. Women victims of IPV will exhibit symptoms of PTSD as indicated by the literature, but will also manifest symptoms of Complex PTSD. There will be a higher prevalence of C-PTSD than PTSD.
3. Neuropsychological alterations in survivor women will be more closely related to specific symptoms of C-PTSD than those of PTSD.
4. The implementation of a neuropsychological rehabilitation program will more effectively improve complex post-traumatic sequelae than classic symptoms.

METHODOLOGY

Design: Randomized controlled trial of parallel groups.

Participants:

Participants:

Participants (objectives 1 and 2):

A total of 100 women victims of IPV (VG group) and 100 non-victimized women (NVG group) aged between 18 and 50 years will be evaluated to avoid age-related deterioration. The women victims included in this study will be randomly selected from the CIMs (Centros de Información a la Mujer) of Andalusia. All participants will sign an informed consent form previously approved by the Committee Ethics Research (CEI Provincial de Granada - A01037775).

Participants (objectives 3 and 4):

The sample will consist of 80 women surivvor of IPV. Among them, 40 will receive neuropsychological rehabilitation program (VIRTRAEL/LUCCIDY) and 40 will receive a standard training for the care of survivor women (TAU), all of the same duration. They will be divided into intervention groups of approximately 6-8 participants (VIRTRAEL/LUCCIDY and TAU). These women will be randomly selected from various CIMs (municipal and provincial) in Andalusia. Inclusion and exclusion criteria will be the same as for the group of survivor women in objectives 1 and 2.

Instruments

Module I: Sociodemographic, clinical, and relationship survey:

* Measures regarding education and socioeconomic level, history of neuropsychological and psychopathological alterations (prior to abuse) that may affect neuropsychological performance (e.g., substance use, medication use, brain diseases, depression, etc.), characteristics of the abusive relationship, time elapsed from the onset of IPV until it was abandoned, among others.
* Alcohol Use Disorders Identification Test-Consumption (Audit-C).

Module II: Variables related to violence:

* World Health Organization violence against women instrument. It is a self-reported questionnaire that assesses the dimensions of physical, sexual, psychological, and, in some versions, economic violence experienced by a woman in the context of Intimate partner violence.
* Adverse Childhood Experiences (ACE). Evaluates exposure to adverse experiences in childhood, including verbal abuse, physical abuse, sexual abuse, among others.
* The International Trauma Exposure Measure (ITEM) is a checklist developed to measure exposure to traumatic life events in a manner consistent with the definition of trauma exposure in the 11th version of the International Classification of Diseases.

Module III: Psychopathological alterations:

* International Trauma Questionnaire (ITQ). Brief self-report measure freely available internationally developed in coherence with ICD-11 criteria (WHO, 2018). It particularly focuses on defining functional impairment for both PTSD and C-PTSD.
* Patient Health Questionnaire (PHQ-9). Evaluates depression through items associated with DSM and ICD criteria. Part of the Patient Health Questionnaire from the National Institutes of Health (NIH).
* Generalized Anxiety Disorder Scale (GAD-7). Screens for generalized anxiety. It has shown solid psychometric properties in the Spanish population, as well as in survivor women of IPV.
* Perceived Stress Scale (PSS). Evaluates perceived stress level and the degree to which individuals find their life unpredictable, uncontrollable, overloaded.
* Emotion Regulation Questionnaire (ERQ). Assesses tendency to regulate emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression.
* Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). It is a self-report questionnaire used to assess PTSD symptoms based on DSM-5 criteria.

Module IV: Neuropsychological assessment:

-BELIEVE Battery. (http://projectbelieve.info). BELIEVE Battery is a free, online and comprehensive neuropsychological battery specifically developed for women victims and survivors of IPV. The Believe Battery includes evidence-based measures for neuropsychological functioning, which were based on the EMBRACED Project. The cognitive domains assessed by this battery include memory, executive function, attention, language, motor and visuospatial abilities, perception, orientation, and social cognition.

Procedure (objectives 3 and 4):

Women will be selected from the population served by different CIMs (Centros de Información a la Mujer) in Andalusia. They will receive detailed information from the research team about the study objectives, as well as the general characteristics of the intervention.

The intervention (VIRTRAEL/LUCCIDY and TAU) will consist of 9 sessions, with a weekly frequency, and in a group format. A psychopathological, DSO, neuropsychological, and previous violence assessment will be conducted (pre and post-treatment and follow-up at 3 months).

The final protocol will adhere to CONSORT criteria, specifically to the recommendations of these criteria for the application to clinical trials of psychological treatments, as well as SPIRIT criteria and its specifications for the consideration of participant self-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write without difficulty.
* For the IPV group, participants must have experienced some form of violence from their partner or ex-partner.

Exclusion Criteria:

* Not having a history of brain damage prior to the abusive relationship
* Not having illnesses prior to the abusive relationship that could affect cognition (e.g., lupus, multiple sclerosis...).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — According to the current legislative framework in Spain, specifically Organic Law 1/2004 on Comprehensive Protection Measures against Gender Violence. This law focuses on violence occurring within the context of intimate partner or ex-partner relationships, where women are the victims of male aggressors.
  However, it is important to highlight that the circumstances and experiences of cisgender women and other women (such as trans women, non-binary individuals, or those of other gender identities) can differ significantly. These differences in the experience of violence and discrimination deserve to be studied separately, as they uniquely affect each group. For example, trans women often face additional barriers in accessing resources and protection, emphasizing the need for an intersectional perspective that addresses the various forms of violence and discrimination experienced by all women.
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological performance | Weeks 2, 15 and 28
  BELIEVE Battery is a computerized battery administered through a tablet that evaluates different cognitive functions: Cancellation measures selective attention; Colored Words assesses flexibility and inhibition; Coin in Hand tests memory under distraction; Visomotor and Alternate Visomotor evaluate processing speed and motor skills; Matrices measures abstract reasoning; Multitasking tests multitasking ability; Working Memory assesses memory with numbers and colors; Verbal Memory tests recall; Verbal Comprehension evaluates instruction understanding; Finger Tapping measures motor speed; Marking, Tracing, Dotting evaluate visuomotor coordination; Complex Figure Copy tests visual memory; Naming tests verbal identification; Fluency tests word generation; Orientation measures awareness; Clock Drawing tests visuoconstruction; Continuous Performance measures attention; Eyes tests emotion recognition; Simple Reaction Time measures motor speed.
Posttraumatic Stress Disorder and Complex-Posttraumatic Stress Disorder | Weeks 1, 14 and 27
  The International Trauma Questionnaire (ITQ) is a tool designed to assess the symptoms of Post-Traumatic Stress Disorder (PTSD) and Complex PTSD as outlined by the International Classification of Diseases.
  Each symptom is rated on a scale from 0 to 4, where: 0 = Not at all; 1 = A little bit; 2 = Moderately; 3 = Quite a bit;4 = Extremely.
  For PTSD, the questionnaire focuses on three core clusters: Re-experiencing the trauma, Avoidance of trauma-related stimuli and Persistent sense of threat or hypervigilance.
  For CPTSD, additional domains are assessed: Affective dysregulation, Negative self-concept and Interpersonal difficulties.
  To meet the criteria for PTSD, the respondent must score at least 2 (moderately) on one symptom from each of the PTSD clusters.
  To meet the criteria for CPTSD, the same PTSD criteria must be met, plus a score of at least 2 on one symptom from each of the disturbances in self-organization (DSO) clusters.

SECONDARY OUTCOMES:
Adverse childhood experiences | Weeks 1, 14 and 27
  Adverse Childhood Experience (ACE). It is a screening tool designed to measure various types of adverse experiences that occur during childhood, such as abuse, neglect, and household dysfunction. The ACE questionnaire consists of 10 questions, each focusing on different types of adverse experiences before the age of 18. The total score, ranging from 0 to 10, indicates the level of exposure to childhood adversity, with higher scores being associated with greater health risks.
Depression | Weeks 1, 14 and 27
  Patient Health Questionnaire (PHQ-9). It is a widely-used self-report tool for assessing depression severity. It consists of 9 items, each of which corresponds to one of the diagnostic criteria for major depressive disorder as outlined in the DSM-IV.
  The PHQ-9 asks individuals to rate the frequency of symptoms such as low mood, loss of interest in activities, changes in sleep and appetite, concentration difficulties, feelings of worthlessness, and thoughts of self-harm over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 27. Higher scores indicate more severe depressive symptoms.
  Scoring guidelines typically classify the severity of depression as:
  0-4: Minimal or none 5-9: Mild 10-14: Moderate 15-19: Moderately severe 20-27: Severe
Anxiety | Weeks 1, 14 and 27
  Generalized Anxiety Disorder Scale (GAD-7). It is a brief self-report tool designed to assess the severity of generalized anxiety disorder (GAD) and anxiety-related symptoms. It consists of 7 items that ask how often, over the last two weeks, the individual has experienced symptoms such as feeling nervous, inability to control worry, restlessness, irritability, and physical symptoms like tension or trouble relaxing.
  Each item is scored from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 21. The higher the score, the more severe the anxiety:
  0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety
Severity and intensity of Intimate partner violence | Weeks 1, 14 y 27
  World Health Organization violence against women instrument. It is a self-reported questionnaire that assesses the dimensions of physical, sexual, psychological, and, in some versions, economic violence experienced by a woman in the context of Intimate partner violence. The response options are typically based on a frequency scale: 0 = never, 1 = once, 2 = a few times, and 3 = many times. To calculate the score, the responses for each dimension of violence are summed, allowing for a measure of the severity and frequency of the violence experienced.
Sociodemographic, clinical, and relationship variables | Weeks 1, 14 and 27
  Measures regarding education and socioeconomic level, history of neuropsychological and psychopathological alterations (prior to abuse) that may affect neuropsychological performance (e.g., substance use, brain diseases, depression, etc.), characteristics of the abusive relationship, time elapsed from the onset of IPV until it was abandoned, among others.
Posttraumatic Stress Disorder | Weeks 1, 14 and 27
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). It is a self-report questionnaire used to assess PTSD symptoms based on DSM-5 criteria. It consists of 20 items covering re-experiencing, avoidance, negative cognition/mood, and hyperarousal symptoms. Responses are rated on a 5-point Likert scale: 0 = Not at all; 1 = A little bit; 2 = Moderately; 3 = Quite a bit; 4 = Extremely The total score is calculated by summing the responses, ranging from 0 to 80, with higher scores indicating greater PTSD symptom severity. A score of 33 or higher is often used as a cut-off for a provisional PTSD diagnosis.
Exposure to traumatic life events | Weeks 1, 14 and 27
  The International Trauma Exposure Measure (ITEM) is a checklist developed to measure exposure to traumatic life events in a manner consistent with the definition of trauma exposure in the 11th version of the International Classification of Diseases. The ITEM measures exposure to 21 different traumatic life events across different developmental periods: childhood, adolescence, and adulthood.
Perceived Stress | Weeks 1, 14 and 27
  Perceived Stress Scale (PSS). It is a tool designed to measure an individuals perception of stress. The PSS assesses perceived stress rather than actual stressors, giving insight into how people interpret and cope with stress in their lives.
  The PSS consists of 10 items that ask about feelings and thoughts during the last month. Respondents rate each item on a 5-point scale ranging from 0 (never) to 4 (very often). Items cover experiences such as feeling nervous or stressed, being able to handle personal problems, and feeling confident about coping with difficulties.
  The total score is calculated by reversing the scores on certain positive items and summing them up, with higher scores indicating higher levels of perceived stress.
Emotion Regulation | Weeks 1, 14 and 27
  Emotion Regulation Questionnaire (ERQ). It is a self-report measure designed to assess individual differences in emotion regulation strategies, particularly focusing on cognitive reappraisal and expressive suppression.
  The ERQ consists of 10 items, with participants rating how often they use these strategies on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Six items assess cognitive reappraisal, and four items assess expressive suppression.
Alcohol Use Disorders | Weeks 1, 14 and 27
  Alcohol Use Disorders Identification Test-Consumption (Audit-C) is a widely used screening tool to identify individuals with risky drinking behaviors and potential alcohol use disorders. the AUDIT-C consists of three questions that assess:
  * Frequency of alcohol consumption (How often do you have a drink containing alcohol?),
  * Quantity of alcohol consumed (How many drinks containing alcohol do you have on a typical day when you are drinking?),
  * Frequency of binge drinking (How often do you have six or more drinks on one occasion?).
  Each question is scored from 0 to 4, with the total score ranging from 0 to 12. Higher scores indicate a greater risk of hazardous drinking or alcohol use disorder. A score of 4 or more in men and 3 or more in women is typically considered positive for identifying hazardous drinking.

CONTACTS AND LOCATIONS:
Locations (1):
- Mind, Brain and Behavior Research Center at University of Granada (CIMCYC-UGR), Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after the identification, will be shared.
  Access Criteria:
  Investigators whose proposed use of the data has been approved by an independent review committee and who provide a methodologically sound proposal. Proposals should be directed to nhidalgo@ugr.es
Supporting Information: Study Protocol, ICF
Time Frame: October 2024-June 2027

REFERENCES:
- [Background] Daugherty, J. C., Marañón-Murcia, M., Hidalgo-Ruzzante, N., Bueso-Izquierdo, N., Jiménez-González, P., Gómez-Medialdea, P., & Pérez-García, M. (2018). Severity of neurocognitive impairment in women who have experienced intimate partner violence in Spain. The Journal of Forensic Psychiatry & Psychology, 30(2), 322-340
- [Background] Cloitre M, Hyland P, Prins A, Shevlin M. The international trauma questionnaire (ITQ) measures reliable and clinically significant treatment-related change in PTSD and complex PTSD. Eur J Psychotraumatol. 2021 Jun 22;12(1):1930961. doi: 10.1080/20008198.2021.1930961. PMID 34211640
- [Background] Fernandez-Fillol C, Pitsiakou C, Perez-Garcia M, Teva I, Hidalgo-Ruzzante N. Complex PTSD in survivors of intimate partner violence: risk factors related to symptoms and diagnoses. Eur J Psychotraumatol. 2021 Dec 16;12(1):2003616. doi: 10.1080/20008198.2021.2003616. eCollection 2021. PMID 34925711
- Available data/document: INFORMATION SHEET — https://drive.google.com/file/d/1Y90Fr8O30tFqNL_OjAjMfrayrK8-KKxt/view?usp=sharing
- Available data/document: Informed Consent Form: Informed Consent Form — https://drive.google.com/file/d/1eQLHRV80sIPlZNoHR5HFS4uauF8RWoDI/view?usp=sharing